CLINICAL TRIAL: NCT03969810
Title: Rounding Summaries for Families of Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Jared Greenberg, Assistant Professor, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19042604
Record Dates: First submitted 2019-05-10; First posted 2019-05-31 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Acute Respiratory Failure; Intensive Care Unit Syndrome; Communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rounding Summary (Experimental): Surrogates who are assigned to the intervention group will receive a written rounding summary every day or every other day that the patient is in the ICU. The summary will be organized as follows for each of the most important ICU problems: 1) Description of the problem, 2) Ways the ICU team is addressing the problem i.e. consultations, diagnostic tests, and treatments. 3) An assessment of whether the problem is improving or worsening.
  For patients assigned to the intervention group, the investigators will forward the previous day's summary to the ICU nurse at the beginning of each day shift. After participating in morning rounds, ICU nurses will be asked to modify the summary based on the plan for the day. Nurses will be asked to use the written summary to guide communication with surrogates that day.
  Interventions: Behavioral: Rounding Summary
- Usual Care (No Intervention): Usual ICU care

INTERVENTIONS:
Behavioral: Rounding Summary — Written summary of rounds
  Arms: Rounding Summary

SUMMARY:
Many patients in intensive care units (ICUs) rely on family members or surrogates to make medical decisions on their behalf. One of the recommended ways to improve a surrogate's experience is to invite him or her to participate in daily, multidisciplinary ICU rounds. In practice, this is often a challenging way for clinicians to engage with the patient's surrogates.

Surrogates of non-decisional ICU patients will be randomized to receive a written rounding summary every day or every other day that the patient is in the ICU. The summary will be organized as follows for each of the most important ICU problems: 1) Description of the problem, 2) Ways the ICU team is addressing the problem i.e. consultations, diagnostic tests, and treatments. 3) An assessment of whether the problem is improving or worsening.

The investigators hypothesize that surrogates who receive written rounding summaries will be more satisfied with ICU care than surrogates who receive usual care. Satisfaction will be measured by the Critical Care Family Needs Inventory (CCFNI) questionnaire.

ELIGIBILITY:
Patients in the adult Medical and Cardiac ICUs at Rush University Medical Center will be prospectively screened.

Inclusion criteria (Patient characteristics required for surrogate inclusion) At least one of the following

* The patient has required invasive or non-invasive mechanical ventilation for at least three consecutive days.
* The patient has an expected in-hospital mortality rate of at least 25% according to the primary ICU physician.

Exclusion criteria (Patient characteristics that will exclude surrogates from study enrollment):

* The patient possesses decisional capacity at the time of enrollment.
* The patient has required invasive or non-invasive mechanical ventilation for more than the previous 14 days
* The patient is expected to die or transition to comfort care within the next 48 hours based on ICU physician estimate.
* The patient is expected to be liberated from mechanical ventilation (if applicable) or discharged from the ICU within the next 24 hours.
* There is no identifiable surrogate.
* The patient is member of a vulnerable population i.e. pregnant, prisoner.
* The ICU physician refuses permission to approach surrogates for consent

The investigators will hand out fliers that describe the study to surrogates of patients who are expected to meet the above criteria. Surrogates can ask the nurse to contact the lead investigator if they are interested in learning more about the study. If no surrogate is present prior to the patient meeting the inclusion criteria, the investigators will attempt to contact the surrogate by phone to provide information on the study.

One surrogate will be approached for informed consent and enrolled based on the following criteria.

Inclusion criteria for surrogate decision maker:

* Age ≥ 18 years old
* Self-identified as participating directly in health care decision making for the incapable patient

Exclusion criteria for surrogate decision makers:

* The surrogate does not agree to participate in study procedures (surveys, interviews)
* The surrogate needs translation assistance because of poor English fluency
* The surrogate has history of a clinically important neurological disorder (e.g., dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-02-12 (Actual)

PRIMARY OUTCOMES:
Surrogate Satisfaction with Patient Care: Critical Care Family Needs Inventory (CCFNI) questionnaire | Measured once 5-7 days after enrollment (or within 24 hours of ICU discharge if this occurs first). For patients who remain in the ICU an additional 5 days after first measurement, the outcome will be measured again.
  Score on the Critical Care Family Needs Inventory (CCFNI) questionnaire. 14 questions. Total score range 14-56 with lower scores indicating better satisfaction.

SECONDARY OUTCOMES:
Surrogate Anxiety and Depression | Measured once 5-7 days after enrollment (or within 24 hours of ICU discharge if this occurs first). For patients who remain in the ICU an additional 5 days after first measurement, the outcome will be measured again.
  Score on Hospital Anxiety and Depression Scale (HADS). Total score 0-21 for anxiety (7 questions) and 0-21 for depression (7 questions). Higher scores indicate greater symptom burden.
Surrogate Symptoms of Post-Traumatic Stress Disorder (PTSD) | Measured once 5-7 days after enrollment (or within 24 hours of ICU discharge if this occurs first). For patients who remain in the ICU an additional 5 days after first measurement, the outcome will be measured again.
  Score on Impact of Events Scale Revised (IES-R) questionnaire. 22 questions. Score 0-88 with higher scores indicating more stress.
Surrogate and physician agreement regarding the patient's condition | Measured once 5-7 days after enrollment (or within 24 hours of ICU discharge if this occurs first). For patients who remain in the ICU an additional 5 days after first measurement, the outcome will be measured again.
  Surrogates and ICU physicians will be provided with a list of common medical ICU diagnoses. Respondents will be asked to indicate which of these diagnoses, if any, pertain to the patient. When the respondent picks a diagnosis, he or she will be prompted to indicate whether common treatments for that condition are being provided. Finally, for each checked diagnosis, the respondent will indicate whether he or she believes the problem is "getting better, getting worse, or staying the same." Members of the research team, blinded to the surrogates' treatment arm, will evaluate for inter-rater agreement between surrogates and ICU physician responses.
Change in Surrogate Satisfaction with Patient Care: Critical Care Family Needs Inventory (CCFNI) questionnaire | From enrollment to 5-7 days after enrollment (or within 24 hours of ICU discharge if this occurs first).
  Change in Score on the Critical Care Family Needs Inventory (CCFNI) questionnaire. 14 questions. Total score range 14-56 with lower scores indicating better satisfaction.
Change in Surrogate Anxiety and Depression | From enrollment to 5-7 days after enrollment (or within 24 hours of ICU discharge if this occurs first).
  Change in Score on Hospital Anxiety and Depression Scale (HADS). Total score 0-21 for anxiety (7 questions) and 0-21 for depression (7 questions). Higher scores indicate greater symptom burden.
Change in Surrogate Symptoms of Post-Traumatic Stress Disorder (PTSD) | From enrollment to 5-7 days after enrollment (or within 24 hours of ICU discharge if this occurs first).
  Change in score on Impact of Events Scale Revised (IES-R) questionnaire. 22 questions. Score 0-88 with higher scores indicating more stress.

OTHER OUTCOMES:
Qualitative feedback from participating surrogates | Measured once 5-7 days after enrollment (or within 24 hours of ICU discharge if this occurs first). For patients who remain in the ICU an additional 5 days after first measurement, the outcome will be measured again.
  All surrogates will be asked to participate in a 10-15 minute phone or in-person interview. This interview will deal with their satisfaction with the patient's care and communication with the ICU staff.
Feedback from participating nurses | Daily while patient is in the ICU
  Nurses of enrolled patients/surrogates will be asked to complete an online survey regarding communication with the patient and/or surrogates that day. Nurses will also be invited to participate in focus groups to provide feedback.
Surrogate Satisfaction with Patient Care | Measured once 10-14 days after enrollment if patient still in ICU
  Score on the Critical Care Family Needs Inventory (CCFNI) questionnaire. 14 questions. Total score range 14-56 with lower scores indicating better satisfaction.
Surrogate Anxiety and Depression | Measured once 10-14 days after enrollment if patient still in ICU
  Score on Hospital Anxiety and Depression Scale (HADS). Total score 0-21 for anxiety (7 questions) and 0-21 for depression (7 questions). Higher scores indicate greater symptom burden.
Surrogate Symptoms of Post-Traumatic Stress Disorder (PTSD) | Measured once 10-14 days after enrollment if patient still in ICU
  Score on Impact of Events Scale Revised (IES-R) questionnaire. 22 questions. Score 0-88 with higher scores indicating more stress.
Surrogate and physician agreement regarding the patient's condition | Measured once 10-14 days after enrollment if patient still in ICU
  Surrogates and ICU physicians will be provided with a list of common medical ICU diagnoses. Respondents will be asked to indicate which of these diagnoses, if any, pertain to the patient. When the respondent picks a diagnosis, he or she will be prompted to indicate whether common treatments for that condition are being provided. Finally, for each checked diagnosis, the respondent will indicate whether he or she believes the problem is "getting better, getting worse, or staying the same." Members of the research team, blinded to the surrogates' treatment arm, will evaluate for inter-rater agreement between surrogates and ICU physician responses.
Patient length of mechanical ventilation (if applicable) | Measured during hospitalization, up to 90 days after enrollment.
  Patient length of mechanical ventilation (if applicable)
Patient failed extubation attempt (yes/no) (if applicable) | Measured during hospitalization, up to 90 days after enrollment.
  Failed extubation attempt (yes/no) (if applicable)
Tracheostomy placement during ICU admission (yes/no) | Measured during hospitalization, up to 90 days after enrollment.
  Tracheostomy placement during ICU admission (yes/no)
Days from intubation to tracheostomy placement (if applicable) | Measured during hospitalization, up to 90 days after enrollment.
  Days from intubation to tracheostomy placement (if applicable)
ICU discharge requiring invasive mechanical ventilation (yes/no) | Measured during hospitalization, up to 90 days after enrollment.
  ICU discharge requiring invasive mechanical ventilation (yes/no)
ICU discharge requiring new artificial nutritional supplementation (yes/no) | Measured during hospitalization, up to 90 days after enrollment.
  ICU discharge requiring new artificial nutritional supplementation (yes/no)
ICU discharge requiring new renal replacement therapy (yes/no) | Measured during hospitalization, up to 90 days after enrollment.
  ICU discharge requiring new renal replacement therapy (yes/no)
Change in code status or limitations to care during ICU stay (yes/no) | Measured during hospitalization, up to 90 days after enrollment.
  Change in code status or limitations to care during ICU stay (yes/no)
Days from ICU admission to change in code status or new limitations to care (if applicable) | Measured during hospitalization, up to 90 days after enrollment.
  Days from ICU admission to change in code status or new limitations to care (if applicable)
ICU length of stay (days) | Measured during hospitalization, up to 90 days after enrollment.
  ICU length of stay (days)
Hospital length of stay (days) | Measured during hospitalization, up to 90 days after enrollment.
  Hospital length of stay (days)
Hospital disposition | Measured during hospitalization, up to 90 days after enrollment.
  Hospital disposition

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Davidson JE, Jones C, Bienvenu OJ. Family response to critical illness: postintensive care syndrome-family. Crit Care Med. 2012 Feb;40(2):618-24. doi: 10.1097/CCM.0b013e318236ebf9. PMID 22080636
- [Background] Nelson JE, Hanson LC, Keller KL, Carson SS, Cox CE, Tulsky JA, White DB, Chai EJ, Weiss SP, Danis M. The Voice of Surrogate Decision-Makers. Family Responses to Prognostic Information in Chronic Critical Illness. Am J Respir Crit Care Med. 2017 Oct 1;196(7):864-872. doi: 10.1164/rccm.201701-0201OC. PMID 28387538
- [Background] Brown SM, Rozenblum R, Aboumatar H, Fagan MB, Milic M, Lee BS, Turner K, Frosch DL. Defining patient and family engagement in the intensive care unit. Am J Respir Crit Care Med. 2015 Feb 1;191(3):358-60. doi: 10.1164/rccm.201410-1936LE. No abstract available. PMID 25635496
- [Background] Davidson JE, Aslakson RA, Long AC, Puntillo KA, Kross EK, Hart J, Cox CE, Wunsch H, Wickline MA, Nunnally ME, Netzer G, Kentish-Barnes N, Sprung CL, Hartog CS, Coombs M, Gerritsen RT, Hopkins RO, Franck LS, Skrobik Y, Kon AA, Scruth EA, Harvey MA, Lewis-Newby M, White DB, Swoboda SM, Cooke CR, Levy MM, Azoulay E, Curtis JR. Guidelines for Family-Centered Care in the Neonatal, Pediatric, and Adult ICU. Crit Care Med. 2017 Jan;45(1):103-128. doi: 10.1097/CCM.0000000000002169. PMID 27984278
- [Derived] Thinnes WE, Harrison MR, Basapur S, Weiss MA, Quinn TV, Ritz EM, Shah RC, Greenberg JA. Written Communication, Visitation Policies, and Awareness of Medical Issues Among Intensive Care Unit Families. Am J Crit Care. 2023 Jul 1;32(4):302-306. doi: 10.4037/ajcc2023986. PMID 37391367
- [Derived] Greenberg JA, Basapur S, Quinn TV, Bulger JL, Schwartz NH, Oh SK, Shah RC, Glover CM. Challenges faced by families of critically ill patients during the first wave of the COVID-19 pandemic. Patient Educ Couns. 2022 Feb;105(2):297-303. doi: 10.1016/j.pec.2021.08.029. Epub 2021 Aug 27. PMID 34507866